CLINICAL TRIAL: NCT00036231
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Multiple Dose Study to Assess the Efficacy, Safety and Tolerability of RG1068 (Synthetic Human Secretin) in Children With Autism and Gastrointestinal Dysfunction
Brief Title: Synthetic Human Secretin in Children With Autism and Gastrointestinal Dysfunction
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Repligen Corporation (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: RG1068-03
Record Dates: First submitted 2002-05-08; First posted 2002-05-09 (Estimated); Last update posted 2005-11-21 (Estimated); Status verified 2005-08

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder | interventions — Secretin

INTERVENTIONS:
Drug: RG1068 (Synthetic Human Secretin)

SUMMARY:
The purpose of the study is to determine the effect of multiple doses of secretin on autism.

ELIGIBILITY:
* Autism
* Gastrointestinal dysfunction

Ages: 32 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2002-04

REFERENCES:
- See also: Related Info — http://www.repligen.com